CLINICAL TRIAL: NCT00442364
Title: An Open Label Multicenter Safety Study of the Varisolve® Procedure for the Treatment of Varicose Veins in Patients With Right-to-left Cardiac Shunt
Brief Title: Safety Study of Varisolve® Procedure for Treatment of Varicose Veins in Patients With Right-to-left Cardiac Shunt
Acronym: MRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAP.VV012
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Varicose Veins
Keywords: PFO; Patent Foramen Ovale; Right-to-Left Shunt; Sclerotherapy
MeSH Terms: conditions — Varicose Veins; Foramen Ovale, Patent | interventions — Polidocanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Polidocanol (1%) Microfoam (Varisolve)
  Interventions: Drug: Polidocanol (1%) Microfoam (Varisolve); Procedure: Endovenous Microfoam Occlusion

INTERVENTIONS:
Drug: Polidocanol (1%) Microfoam (Varisolve) — Varisolve polidocanol 1% microfoam, maximum of 20ml injected into affected great saphenous vein.
Procedure: Endovenous Microfoam Occlusion — Varisolve® polidocanol microfoam injection under duplex guidance to fill proximal and distal great saphenous vein and varicose tributaries.

SUMMARY:
The purpose of this study is to determine the safety of the Varisolve® procedure in patients with right-to-left cardiac shunt (a defect in the heart).

DETAILED DESCRIPTION:
Varicose veins are extremely common, affecting up to 25% of the western adult population. While in their early stages they are little more than a sometimes-painful aesthetic problem, progression is inevitable and some will progress to more severe and largely irreversible problems of chronic venous insufficiency (CVI) and, finally, venous leg ulcer. At present, no system has been proven to identify those that will progress and while varicose veins are not the only cause of CVI, in approximately 50% of patients with leg ulcers, superficial varicose veins are the only causal factor identified. The cost of management of simple varicose veins is relatively small in comparison with the long-term management of CVI and leg ulcers. Many patients progress to develop leg ulcers without having received primary treatment for their varicose veins.

The current management of major varicose veins includes maintenance by compression stockings, injection sclerotherapy with liquid sclerosants, and superficial vein surgery. The disadvantages to surgery include the use of general anesthesia, incisions resulting in possible scars, a painful recovery period with significant functional down time and historically high rates of recurrence. Sclerotherapy has been performed since 1851 with the advent of hypodermic needles. The two surfactant sclerosants most widely used are sodium tetradecyl sulphate (STS, STD®, Sotradecol or Fibro-vein) and polidocanol (Macrogol 400 Ph Eur, Aethoxyskerol®). Sotradecol is the only FDA-approved sclerosant. With the advent of duplex ultrasound scanning, the technique of echo-guided sclerotherapy has widened the possibilities for sclerotherapy of large veins but the liquid sclerosants available are rapidly deactivated and diluted by blood frequently resulting in unsatisfactory outcomes. Because the microfoam delivers sclerosant more efficiently to the venous endothelium, it is believed that lower concentrations of polidocanol (Varisolve)can be used when compared with liquid sclerosant. BTG International Ltd is developing sclerosant microfoam technology based on polidocanol (PD)(Varisolve) into a pharmaceutical product.

The presence of bubbles in the heart has been a concern as bubbles may pass from the right heart to the left through a patent foramen ovale (PFO) or other right-to-left shunt. Once in the systemic circulation, some bubbles inevitably pass into the cerebral circulation where their theoretical potential for causing damage due to occlusion of vessels is recognized yet ill defined.

Therefore this study is to determine whether patients with bubbles detected in the middle cerebral artery (MCA) during the Varisolve® procedure experience any sub-clinical, safety-related events such as abnormalities on brain MRI, neurological examination, cardiac markers or other symptoms or signs.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 60 with severe varicose veins, CEAP classes 3, 4 and 5 (CEAP is a classification and grading system for chronic venous disease)
* Saphenofemoral junction (SFJ) incompetence. Retrograde blood flow in the GSV, greater than or equal to 1.0 second demonstrated by duplex scanning.
* Normal MRI, as assessed on MRI examination performed within 5 days prior to procedure.
* Patient must be willing and able to participate in the study and provide written informed consent.

Exclusion Criteria:

* Presence of venous ulcers (i.e. CEAP classification C6) or local infection in the limb to be treated.
* Incompetence of the small saphenous vein (SSV) in the leg to be treated. Venographic or ultrasonographic evidence of current or previous deep vein thrombosis (DVT) (see Appendix IV).
* Deep venous occlusion and/or incompetence. Evidence of deep venous reflux is acceptable if it is confined to a limited segment caused by filling of the incompetent superficial system through a perforator or the SFJ.
* Patients with known atherosclerotic disease or presence of major risk factors, including LDL cholesterol greater than 130 mg/dl, blood pressure greater than 140 mmHg systolic or 90 mmHg diastolic, or diabetes requiring treatment with oral hypoglycemic drugs or insulin.
* Smokers.
* History suggestive of cerebral atherosclerosis, transient ischemic attack (TIA), stroke, presence of carotid bruit or history of abnormal carotid duplex examination.
* Clinically significant dilated cardiomyopathy, evidence of regional wall motion abnormalities suggestive of prior myocardial infarction, rheumatic mitral valve disease, moderately severe or worsening cardiac valvular disease (> 2+ on a scale of 4), known or suspected congenital heart disease, evidence of right sided volume or pressure overload, history of atrial fibrillation. Patients with PFO, atrial septal defect, or other right-to-left shunt are not excluded unless associated with other abnormalities as above.
* Peripheral vascular disease.
* Spontaneous emboli seen on TCD prior to contrast injection.
* Body Mass Index >30.0.
* Recent or current upper respiratory tract illness or other cause of increased coughing.
* Arterial insufficiency in the leg to be treated (ankle: brachial pressure ratio less than 0.9).
* Reduced mobility - unable to maintain a brisk walk unaided for a minimum of 5 minutes per hour per day.
* Prolonged automobile or air travel (>4 hours) 1 month prior to treatment, or planned within 1 month of proposed treatment.
* Current or prior pulmonary embolism.
* Major surgery, prolonged hospitalization or pregnancy within 3 months of screening.
* Hormone replacement therapy or hormonal contraception (oral or dermal patch).
* Current or recent (<7 days before treatment) aldehyde dehydrogenase inhibitor therapy, e.g. disulfiram, or other drugs with similar reactions to alcohol (metronidazole, tinidazole).
* Current anticoagulation therapy.
* Inability to identify a unilateral or bilateral temporal bone window and middle cerebral artery signal by transcranial Doppler ultrasound.
* Inability to undergo magnetic resonance imaging of the brain
* Participation in a clinical study involving an unlicensed pharmaceutical product within the 3 months of screening.
* Previous enrollment in this study.
* Major co-existing disease (e.g. malignancy, pulmonary disease, renal or hepatic insufficiency).
* Known allergic response to polidocanol or severe and multiple allergic reactions.
* Women of childbearing potential not using effective contraception
* Pregnant or lactating women.
* Current alcohol or drug abuse.
* Clinically significant laboratory abnormalities in the opinion of the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Rush, MD, Study Director — BTG International Inc.
Locations (7):
- United States (7):
  - Los Angeles, California
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Polidocanol 1% Injectable Microfoam: polidocanol injectable microfoam 1%
Period: Overall Study
Arm/Group | Polidocanol 1% Injectable Microfoam
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with bubbles detected on MRI
Groups:
- Safety Evaluable: patients treated with polidocanol 1% injectable foam with circulating bubbles present on MRI
Arm/Group | Safety Evaluable
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 59
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Patients With Circulating MCA Bubbles Present on MRI Who Had Signficant Clinical or Neurological Effects
Time Frame: 28 day followup
Measure: Number; unit: participants
Groups:
- Safety Evaluable Population: polidocanol injectable foam 1% with circulating MCA bubbles present at MRI
Arm/Group | Safety Evaluable Population
Number analyzed (Participants) | 60
participants | 0

ADVERSE EVENTS:
Time Frame: 12 months after treatment
Arm/Group | Safety Evaluable
Serious Adverse Events (participants affected / at risk) | 4/60
Other Adverse Events (participants affected / at risk) | 30/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Evaluable (N=60)
Deep vein thrombosis (Vascular disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Evaluable (N=60)
Pain in extrermity (General disorders) | 24 (24)
hematoma evacuation (Vascular disorders) | 8 (8)
deep vein thrombosis (Vascular disorders) | 3 (3)
limb discomfort (Musculoskeletal and connective tissue disorders) | 3 (3)
ecchymosis (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No